CLINICAL TRIAL: NCT02060227
Title: Approach to Shoulder Instability: a Randomized, Controlled Trial
Brief Title: Approach to Shoulder Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20130704-01H
Record Dates: First submitted 2014-01-21; First posted 2014-02-12 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Anterior Shoulder Instability
Keywords: Latarjet; Bankart

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic Bankart repair (Active Comparator): After the diagnostic arthroscopy is completed, any other pathology is documented. At least 3 anchors will be used for the bankart repair for repair of the labrum with an inferior to superior capsular shift. The suture anchors used will be at the discretion of the surgeon but will be of the screw-in variety. The sutures are passed through the labrum, and the labrum is tied to the glenoid rim after the bone is prepared in the standard fashion. The surgical times will be recorded on standardized forms.
  Interventions: Procedure: Arthroscopic Bankart repair
- Open Latarjet procedure (Active Comparator): A deltopectoral approach is used. The coracoacromial ligament (CAL) is exposed and incised 1 cm from its coracoid attachment. Harvesting of a 2.5- to 3-cm coracoid graft allows use of 2 screws for fixation to the glenoid neck through a subscapularis-splitting approach. The stump of the CAL is repaired to the capsule with the arm positioned in neutral. The graft is placed in a extra-articular fashion with capsular closure to the native glenoid rim.
  Interventions: Procedure: Open Latarjet procedure

INTERVENTIONS:
Procedure: Open Latarjet procedure
  Arms: Open Latarjet procedure
Procedure: Arthroscopic Bankart repair
  Arms: Arthroscopic Bankart repair

SUMMARY:
The primary research question is to determine whether patients who undergo a stabilization of the shoulder using a novel decision-making algorithm (ISIS Score) have improved disease-specific quality of life at 1 year post-operatively, as measured by the Western Ontario Instability Index (WOSI) compared with patients who undergo stabilization using a conventional decision-making algorithm. Secondary outcomes include the American Shoulder and Elbow Surgeon's (ASES) score, and difference in recurrence rates of dislocation between the two decision-making algorithms.

DETAILED DESCRIPTION:
The bony architecture of the glenohumeral joint is often likened to that of a golf ball and tee. This geometry provides a functional benefit by allowing for a large arc of motion, but also confers an inherent instability that can result in traumatic anterior shoulder dislocation. By far the most common type of glenohumeral instability is anterior dislocation, accounting for over 90% of all shoulder dislocations. The glenohumeral joint relies on a complex network of static and dynamic structures that aid in stabilizing the joint. Compromise of these structures leads to dislocation and often, recurrent instability. Structures providing static stability to the glenohumeral joint include the congruency of the humeral head and glenoid, the glenoid labrum, glenohumeral ligaments surrounding the joint, and negative intra-articular pressure. Dynamic stabilizers are primarily muscular and include the rotator cuff, which provides a compressive stabilizing effect, the tendon of the long head of the biceps, and muscles that stabilize the scapula.

The current accepted "standard" protocol depends on the amount of glenoid bone loss. Typically, when there is little bone loss, the treatment of anterior recurrent instability involves Bankart arthroscopic stabilization. In the setting of significant glenoid bone loss (>25%), the Latarjet technique involving bone grafting of the glenoid defect is indicated in order to address the aforementioned higher risk of recurrence in this setting.

Balg and Boileau proposed a comprehensive score in 2007 including: age at surgery, degree of sport participation (pre-operative), type of sport (pre-operative), shoulder hyperlaxity, Hill-Sachs on AP radiograph and glenoid loss of contour on AP radiograph at the first consultation: the Instability Severity Index Score (ISIS). In contrast to the standard treatment protocol, the authors propose that an ISIS ≦3 points is an indication for arthroscopic Bankart repair, and a score of greater than 3 is an indication for a Latarjet procedure (open stabilization with coracoid bone graft).

This study would be the first to investigate the ISIS decision-making algorithm, an exciting and novel approach to the treatment of shoulder instability, and to compare it to the conventional treatment algorithm within the framework of a prospective, randomized controlled study. If the new ISIS decision-making algorithm proves to be effective at decreasing recurrence instability rates, improving function and quality of life, while maintaining low complication rates, it has the potential to lead to widespread practice change within the Orthopaedic community in North America and abroad.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent anterior instability (dislocation or subluxation) with or without hyperlaxity, including a clinical history of traumatic anterior instability of the shoulder, with positive apprehension or relocation tests.
2. Provide consent

Exclusion Criteria:

1. Patients with a concomitant rotator cuff lesion or humeral avulsion of the anteroinferior glenohumeral ligament (HAGL)
2. An acute first-time dislocation
3. Previous shoulder surgery
4. Surgery for a painful, unstable shoulder without true dislocation or subluxation
5. Patients with active worker's compensation claims (due to the expectation of lower rates of success in this patient population)
6. Active joint or systemic infection
7. Patients with convulsive disorders, collagen diseases, previous shoulder surgeries, and any other conditions that might affect the mobility of the joint
8. Major medical illness (life expectancy less than 2 years or unacceptably high operative risk)
9. Unable to speak or read English/French
10. Inability to provide informed consent and comply with requirements of participation
11. Unwilling to be followed for 2 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Shoulder Instability Index (WOSI) | From baseline to up until 24-Months Post-Operative
  The Western Ontario Shoulder Instability Index (WOSI) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WOSI is a patient-reported measure, 21-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.

SECONDARY OUTCOMES:
Change in The American Shoulder and Elbow Surgeon's (ASES) | From baseline to up until 24-Months Post-Operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Change in Arthritis Progression | From baseline to up until 24-Months Post-Operative
  Radiological parameters will be examined using x-rays. These images will be analyzed for abnormalities by a Musculoskeletal Radiologist. Higher abnormality incidence indicates worse outcomes.
Adverse Events | From time of enrollment up until 2-years post-operative
  Rates of study adverse events or serious adverse events (e.g. number of re-operations) will be monitored and recorded and compared between study groups. A higher rate of adverse events indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - Pan Am Clinic Foundation, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No